CLINICAL TRIAL: NCT06544967
Title: Sexual Dimorphism of The Fetal Brain Biometry: An Ultrasound-Based Study
Brief Title: Differences Between Male and Femal Fetal Brain Biometry by Ultrasound
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abdelrhman Fathy Mahmoud, Obestitric and Gynecology specialist, Sohag University
Other Study IDs: Soh-Med-24-05-05MD
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Fetal Brain Biometry by Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Male fetuses between 18 to 36 weeks: Ultrasound biometry
- Female fetuses between 18 to 36 weeks: Ultrasound biometry

SUMMARY:
Differences of fetal brain biometry as Biparietal diameter,Head circumference,Transcerebellar diameter, Cavum septum pellucidum as regard to fetal gender by ultrasound

ELIGIBILITY:
Inclusion Criteria:

* healthy women from 18 to 36 weeks gestation of pregnant cases aged from 18 to 40 years normal body mass index range from 18 to 25

Exclusion Criteria:

* Pregnant women with any chronic or systemic disease and fetuses with chromosome anomalies or developmental retardation were not included in the study

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: healthy women from 18 to 36 weeks gestation of pregnant cases aged from 18 to 40 years normal body mass index range from 18 to 25
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Fetal brain biometry | 6 months
  In male and female fetuses

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt